CLINICAL TRIAL: NCT05376930
Title: A Multi-center, Open-label, Extension Study to Evaluate the Long-term Safety and Efficacy of DWP16001 in Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Evaluate the Long Term Safety and Efficacy of DWP16001 Compared to Placebo in the Treatment of T2DM.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001301_Ext
Record Dates: First submitted 2022-01-09; First posted 2022-05-17 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-01

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DWP16001 (Experimental): DWP16001 Tablets
  Interventions: Drug: DWP16001 Amg

INTERVENTIONS:
Drug: DWP16001 Amg — DWP16001 Amg, Tablets, Orally, Once daily

SUMMARY:
The purpose of this study is evaluate the long term safety and efficacy of DWP16001 compared to placebo in the treatment of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in the prior phase 3 study (Protocol No: DW_DWP16001301) for meeting the inclusion criteria and completed the study
2. Voluntarily decided to participate in the extension study and provided a written consent on the consent form

Exclusion Criteria:

1. Those who dropped out of the previously conducted phase 3 clinical trial (Protocol No: DW_DWP16001301)
2. Pregnant or lactating women or those who do not consent to the use of appropriate contraceptive methods during clinical trials Appropriate method of birth control for you or your partner: You must agree to one of the following

   * Either surgical sterilization (vasectomy, etc.) or insertion of an intrauterine device (copper loop, intrauterine hormone-containing system), or
   * A physical barrier method combined with either systemic hormonal contraceptives or spermicide, or
   * Use of male condom combined with either cervical cap or diaphragm
3. In case the investigator judges that participation in this extended clinical trial is inappropriate in consideration of the 24-week observation progress in the previously conducted phase 3 clinical trial (Protocol No: DW_DWP16001301)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Adverse events (AEs) and adverse events of special interest (AESIs)* at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  *Hypoglycemia, urinary tract infection, genital infection, pollakiuria, or polyuria

SECONDARY OUTCOMES:
Changes from baseline* in HbA1c at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  * Visit 2 (randomization) of the prior phase 3 study (Protocol No: DW_DWP16001301)
Changes from baseline* in FPG at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  * Visit 2 (randomization) of the prior phase 3 study (Protocol No: DW_DWP16001301)
Proportion of subjects achieving HbA1c target of < 7% at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP | at Weeks 6, 12, 18, 24, 38, and 52 after administration of the IP
  * Visit 2 (randomization) of the prior phase 3 study (Protocol No: DW_DWP16001301)

CONTACTS AND LOCATIONS:
Locations (1):
- Daewoong pharmatceutical, Seoul, South Korea